CLINICAL TRIAL: NCT03210532
Title: Evaluate the Efficacy and Safety of Combination Treatment With DW1501-R1+DW1501-R2 Versus DW1501-R1 or DW1501-R2+DW1501-R3 in Patients With Hypertension and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1501-301
Record Dates: First submitted 2016-10-12; First posted 2017-07-07 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Telmisartan; Amlodipine; Rosuvastatin Calcium; telmisartan amlodipine combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Test (Experimental): qd PO, Twynsta(telmisartan/amlodipine) + Crestor(rosuvastatin)
  Interventions: Drug: Telmisartan + Amlodipine + Rosuvastatin
- Reference 1 (Active Comparator): qd PO, Micardis(telmisartan) + Crestor(rosuvastatin)
  Interventions: Drug: Telmisartan + Rosuvastatin
- Reference 2 (Active Comparator): qd PO,Twynsta(telmisartan/amlodipine)
  Interventions: Drug: Telmisartan + Amlodipine

INTERVENTIONS:
Drug: Telmisartan + Amlodipine + Rosuvastatin — Telmisartan + Amlodipine + Rosuvastatin + Telmisartan placebo
  Arms: Test
Drug: Telmisartan + Amlodipine — Telmisartan + Amlodipine + Rosuvastatin placebo + Telmisartan placebo
  Arms: Reference 2
Drug: Telmisartan + Rosuvastatin — Telmisartan + Amlodipine placebo + Rosuvastatin + Telmisartan placebo
  Arms: Reference 1

SUMMARY:
A Multicenter, Randomized, Double-blinded, Double-dummy, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Combination Treatment with DW1501-R1+DW1501-R2 Versus DW1501-R1 or DW1501-R2+DW1501-R3 in Patients with Hypertension and Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Adults both male and female who are ≥19,<80 years old
* at screening, 140mmHg≤ SBP<180mmHg & 90mmHg≤ DBP<110mmHg & LDL-C≤250mg/dL & triglyceride<400mg/dL

Exclusion Criteria:

* at screening, the difference BP of one-side arm is SBP ≥ 20mmHg and DBP ≥ 10mmHg
* secondary hypertension or secondary dyslipidemia
* patients who have uncontrolled diabetes melitus, hyper/hypothyroidism or cardiac disease
* women who are pregnant or lactating

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change of MSSBP(Mean Sit Systolic Blood Pressure) from baseline | 8-week
Change of LDL-C(Low Density Lipid Cholesterol) from baseline | 8-week

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance Hospital, Seoul, South Korea